CLINICAL TRIAL: NCT05744206
Title: Validation of Electrocardiogram Waveform, Heart Rate Accuracy and Arrhythmia Diagnosis Concordance in Patients With Cardiac Arrhythmia Using Single-channel ECG Monitoring Patch and Holter Monitoring
Brief Title: Validation of ECG Waveform and Arrhythmia Diagnosis Concordance Using ECG Monitoring Patch and Holter Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mezoo Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDV-2022-01
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Arrhythmias, Cardiac
Keywords: ECG monitoring patch; Validation of Electrocardiogram waveform; Validation of heart rate accuracy; Validation of arrhythmia diagnosis concordance; Patients with cardiac arrhythmia; Holter; Wearable patch-type electrocardiograph
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrocardiogram measurements by holter device and patch-type electrocardiographic at the same time (Experimental): The patient is measured electrocardiogram simultaneously through a holter device and patch-type electrocardiograph
  Interventions: Other: Electrocardiogram measurements by holter device and patch-type electrocardiographic at the same time

INTERVENTIONS:
Other: Electrocardiogram measurements by holter device and patch-type electrocardiographic at the same time — The patient is measured electrocardiogram simultaneously through a holter device and patch-type electrocardiograph

SUMMARY:
This study will verify the 1-channel patch-type ECG's arrhythmia diagnostic concordance rate and electrocardiogram measurement performance by collecting ECG signals from patch-type ECG and Holter device simultaneously for data analysis.

DETAILED DESCRIPTION:
[How to conduct research] This study targeted adults aged 19 years or older. Written consent is obtained from those who are diagnosed with arrhythmia and need a Holter examination among outpatients or inpatients at the Cardiology Department of Kosin University Gospel Hospital. The medical staff attaches the Holter device to the subject and the patch-type electrocardiograph in the Holter examination room. Holter device and patch-type electrocardiograph are returned to the Holter examination room after measuring the electrocardiogram for 24 hours. ECG signals from patch-type electrocardiographs and commercial Holter device and arrhythmia detection information are compared and analyzed.

[Number of Subjects] The number of this study is 105. Written consent is obtained from those who are diagnosed with arrhythmia and need a Holter examination among outpatients or inpatients at the Cardiology Department.

[Data analysis plan] In this study, the personal identification information of the subjects will be coded non-identifying and the collected electrocardiogram data will be stored in the cloud with restricted access from outsiders. Coded, non-identified research data is stored and managed in the cloud in compliance with privacy standards and information security standards. ECG data transmitted through the mobile application is stored in the cloud. Confidentiality and security of data are guaranteed, and data collected from patch-type electrocardiograph is used only for research. The electrocardiogram data acquired in this study are obtained in TXT or MAT format and used for data analysis.

The efficacy evaluation items are as follows.

1. Comparison of ECG signal concordance
2. Comparison of the parameters below for a noise-free section of about 1 minute, not the entire section

   * P-wave, QRS-complex, T-wave: Sensitivity, Positive Predictive Value, Amplitude difference, Correlation to the entire signal
   * P, QRS, T (On/Off time): Time difference
   * PR, QRS, QT (Duration/Interval): Time difference
3. Comparison of arrhythmia diagnosis concordance rates between 24-hour patch-type electrocardiograph and commercial Holter device measurement data by arrhythmia categories (total of 19 including ventricular ectopic beat)

The evaluation method and interpretation method are as follows.

1. In the case of categorical variables, the sensitivity and positive predictive value are evaluated, and in the case of continuous variables, the concordance between the measured values measured by the patch-type electrocardiograph and the Holter device is evaluated using the Bland-Altman plot.
2. Amplitude difference of P-wave, QRS-complex and T-wave & Correlation to the entire signal

   * Peaks of P-wave, QRS-complex (R-wave peaks) and peaks of T-wave are manually annotated in the holter device and patch-type ECG independently to assess amplitude difference and correlation to the entire ECG signal.
3. Time difference of P, QRS, T (On/Off time) & PR, QRS, QT (Duration/Interval)

   * Exact timing of fiducial markers such as onset of P-wave and QRS-complex, and offset of P-wave, QRS-complex, T-wave and clinically useful intervals and durations (PR-interval, RR interval, QT interval, P-wave duration, QRS-duration) are manually annotated in the holter device and patch-type ECG independently to quantify the accuracy of delineating these characteristic points in the patch sensor.
4. Root Mean Square of Heart Rate

   * Calculate and analyze the square root after averaging the squares of each heart rate value in the analysis section from the electrocardiogram obtained simultaneously from the Holter device and the patch-type electrocardiograph

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years of age or older
* Patients who are diagnosed with arrhythmia and need regular Holter electrocardiography among outpatients or hospitalized patients at the Department of Cardiology, Kosin University Gospel Hospital
* Those who gave written consent to this clinical study
* Able to understand and carry out training and instructions

Exclusion Criteria:

* A person with a physical disability that cannot wear a patch-type electrocardiograph
* A person suffering from skin disease or functional disorder at the site where the patch-type electrocardiograph will be attached
* Subjects who cannot read the consent form (illiterate, foreigners, etc.)
* Patients judged to be unsuitable for participation in this clinical study by the judgment of investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of arrhythmia diagnosis concordance rates between patch-type electrocardiograph and commercial Holter device measurement data by arrhythmia categories | Within 3 months after electrocardiogram procedure
  Comparison of arrhythmia diagnosis concordance rates between 24-hour patch-type electrocardiograph and commercial Holter device measurement data by arrhythmia categories(total of 19 including ventricular ectopic beat)
Comparison of ECG signal concordance between patch-type electrocardiograph and holter device | Within 3 months after electrocardiogram procedure
  Calculate the concordance (%) of the ECG signal by comparing and analyzing total QRS complex, total ventricular ectopic beat, total atrial ectopic beats, minimum heart rate, maximum heart rate, average heart rate and maximum RR interval

CONTACTS AND LOCATIONS:
Overall Officials: JH Park, Study Director — CEO
Locations (1):
- Kosin University Gospel Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajbhandary PL, Nallathambi G, Selvaraj N, Tran T, Colliou O. ECG Signal Quality Assessments of a Small Bipolar Single-Lead Wearable Patch Sensor. Cardiovasc Eng Technol. 2022 Oct;13(5):783-796. doi: 10.1007/s13239-022-00617-3. Epub 2022 Mar 15. PMID 35292914
- [Background] Yenikomshian M, Jarvis J, Patton C, Yee C, Mortimer R, Birnbaum H, Topash M. Cardiac arrhythmia detection outcomes among patients monitored with the Zio patch system: a systematic literature review. Curr Med Res Opin. 2019 Oct;35(10):1659-1670. doi: 10.1080/03007995.2019.1610370. Epub 2019 May 28. PMID 31045463
- [Background] Fung E, Jarvelin MR, Doshi RN, Shinbane JS, Carlson SK, Grazette LP, Chang PM, Sangha RS, Huikuri HV, Peters NS. Electrocardiographic patch devices and contemporary wireless cardiac monitoring. Front Physiol. 2015 May 27;6:149. doi: 10.3389/fphys.2015.00149. eCollection 2015. PMID 26074823
- [Background] Liu CM, Chang SL, Yeh YH, Chung FP, Hu YF, Chou CC, Hung KC, Chang PC, Liao JN, Chan YH, Lo LW, Wu LS, Lin YJ, Wen MS, Chen SA. Enhanced detection of cardiac arrhythmias utilizing 14-day continuous ECG patch monitoring. Int J Cardiol. 2021 Jun 1;332:78-84. doi: 10.1016/j.ijcard.2021.03.015. Epub 2021 Mar 13. PMID 33727122
- [Background] Solomon MD, Yang J, Sung SH, Livingston ML, Sarlas G, Lenane JC, Go AS. Incidence and timing of potentially high-risk arrhythmias detected through long term continuous ambulatory electrocardiographic monitoring. BMC Cardiovasc Disord. 2016 Feb 17;16:35. doi: 10.1186/s12872-016-0210-x. PMID 26883019
- [Background] Kancharla K, Estes NAM. Mobile cardiac monitoring during the COVID-19 pandemic: Necessity is the mother of invention. J Cardiovasc Electrophysiol. 2020 Nov;31(11):2812-2813. doi: 10.1111/jce.14726. Epub 2020 Sep 3. No abstract available. PMID 32852854
- [Background] Xia H, Garcia GA, Zhao X. Automatic detection of ECG electrode misplacement: a tale of two algorithms. Physiol Meas. 2012 Sep;33(9):1549-61. doi: 10.1088/0967-3334/33/9/1549. Epub 2012 Aug 17. PMID 22903067
- [Background] Krahn AD, Klein GJ, Yee R, Skanes AC. Detection of asymptomatic arrhythmias in unexplained syncope. Am Heart J. 2004 Aug;148(2):326-32. doi: 10.1016/j.ahj.2004.01.024. PMID 15309004